CLINICAL TRIAL: NCT03876353
Title: Efficacy of Flossing in the Removal of Oral Plaque Biofilm
Brief Title: University of New Mexico Dental Hygiene
Acronym: UNM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Lindsey Lee, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 17-419
Record Dates: First submitted 2019-02-26; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Oral Plaque Biofilm
MeSH Terms: interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Side (Other): Each participant who participate will have half of their mouth flossed. Either the right or the left side. The investigator will not know which side has been flossed prior to documenting any tooth surfaces with residual plaque
  Interventions: Other: Floss
- Right Side (Other): Each participant who participate will have half of their mouth flossed. Either the right or the left side. The investigator will not know which side has been flossed prior to documenting any tooth surfaces with residual plaque
  Interventions: Other: Floss

INTERVENTIONS:
Other: Floss — All participants will have half of their mouth flossed. Each participant will act as their own control.

SUMMARY:
To evaluate the efficacy of flossing in the removal of oral plaque biofilm.

DETAILED DESCRIPTION:
Flossing is universally recognized in the dental profession as a primary component of oral hygiene. Data supports the correlation between flossing and disease prevention by ways of reducing gingival bleeding, gingivitis, and dental caries.(1, 2) However, a recent AP publication (3) questioning the validity of flossing as an efficacious preventative method has warranted that oral healthcare professionals address certain underlying assumptions about the practice. Specifically, there is a clear gap in the number of clinical effectiveness trials that measure the ability of flossing for the sole purpose of oral plaque biofilm removal. Such studies are urgently needed. At this moment we can only assume flossing's correlation with disease prevention also links flossing with effectively removing oral plaque biofilm. Due to the current research gaps, additional studies must be performed to address the needs highlighted by the absence of substantive research in this field.

Our long term goal is to evaluate if flossing is an effective oral health aid in the removal of oral plaque biofilm. The overall objective of this application is to provide a consistent measurement to confirm whether flossing is an effective oral care technique in removing disease causing oral plaque biofilm . The rationale that underlies this proposal comes from the many professional associations, such as the American Dental Association, American Dental Hygienists' Association, and the U.S. Department of Health and Human Services, that endorse flossing as an effective home care routine in oral disease prevention. Many oral health professionals would argue that flossing is effective in plaque removal, as they have seen the results anecdotally year after year, yet it is clear that additional studies are needed to move what is known anecdotally to what is known scientifically.

ELIGIBILITY:
Inclusion Criteria:

* Any persons 18 years of age and able to consent

Exclusion Criteria:

A person being edentulous or who have teeth that do not contact Allergy to erythrosine dye (red #3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
measure removal of oral plaque biofilm | 15 minutes
  Evaluate the correlation between flossing and oral plaque biofilm formation

CONTACTS AND LOCATIONS:
Locations (1):
- Universsity of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No